CLINICAL TRIAL: NCT01072838
Title: Safety and Feasibility of Short-Course, Accelerated, Hypofractionated Partial Breast Radiotherapy in Women With Early Stage Breast Cancer Using the Contura MLB Breast Brachytherapy Catheter: A Phase II Trial
Brief Title: Safety Study for Short-course Accelerated, Hypofractionated Partial Breast Radiotherapy (APBI) in Women With Early Stage Breast Cancer Using the Contura MLB
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: SenoRx, Inc. (Industry)
Collaborators: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S09-001; NCT01019720 (obsolete NCT alias)
Record Dates: First submitted 2010-02-18; First posted 2010-02-22 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; APBI; brachytherapy; Contura
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose Escalation (Other)
  Interventions: Radiation: APBI (Dose Escalation); Device: Contura MLB Breast Brachytherapy Catheter

INTERVENTIONS:
Radiation: APBI (Dose Escalation) — Accelerated, hypofractionated partial breast radiotherapy.
  3 dose schemes followed for 6 months each.
Device: Contura MLB Breast Brachytherapy Catheter

SUMMARY:
To determine local disease control (recurrence) with shorter course of APBI delivered with a breast brachytherapy applicator.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy > 10 years
* Lumpectomy with clear margins (negative per NSABP criteria)
* DCIS and/or invasive carcinoma
* If invasive, nodes must be negative
* T stage is Tis, T1 or T2<=3 cm max diameter
* ER(+) or ER(-)/PR(+)

Exclusion Criteria:

* Pregnant or breast feeding
* Active collagen-vascular disease
* Paget's disease of the breast
* Prior history of breast cancer
* Prior breast or thoracic radiotherapy
* Multicentric carcinoma
* Synchronous bilateral breast cancer
* Surgical margins that cannot be assessed or that are positive
* T Stage is T2>3 cm or greater
* ER(-)/PR(-)

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Delivery of short-course APBI will result in locoregional disease control that is equal to that reported for conventional fractionation schemes for APBI. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Atif Khan, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey; Douglas W. Arthur, MD, Principal Investigator — Virginia Commonwealth University; Mihai Ghilezan, MD, Principal Investigator — Corewell Health East
Locations (3):
- United States (3):
  - William Beaumont Hospital, Royal Oak, Michigan
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Virginia Commonwealth University, Richmond, Virginia